CLINICAL TRIAL: NCT02837653
Title: Efficacy of a Physical Activity Counselling on the Severity of Chronic Low Back Pain in Patients With Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEULS-PI-108/2016
Record Dates: First submitted 2016-06-29; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Low Back Pain; Physical Activity
Keywords: cardiovascular Risk
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental (Experimental): Usual Care in Primary Health Care in Low back pain patients, consisting in Therapeutic Exercise and Superficial Thermotherapy at home, and a personalized Physical Activity Counseling based on the Cardiovascular Risk of Each Patient
  Interventions: Behavioral: Physical Activity Counselling; Other: Therapeutic Exercise for LBP; Other: Superficial Thermotherapy
- Control (Active Comparator): Usual Care in Primary Health Care in Low back pain patients, consisting in Therapeutic Exercise and Superficial Thermotherapy at home.
  Interventions: Other: Therapeutic Exercise for LBP; Other: Superficial Thermotherapy

INTERVENTIONS:
Behavioral: Physical Activity Counselling
  Other Names: Physical Activity Advice
  Arms: Experimental
Other: Therapeutic Exercise for LBP
Other: Superficial Thermotherapy

SUMMARY:
Objective: To determine the influence of a counseling of physical activity (PA) versus usual care (UC) in the magnitude of chronic pain (CP) in patients diagnosed with chronic low back pain (CLBP).

Methods: A total of 64 subjects with (CLBP) and older were randomly divided into two groups: an experimental group (UC) + counseling of (AF) and control group (UC). Each group consisted of 32 participants and were evaluated twice (pre and post-intervention), being spaced one month, both groups received telephone follow-up for their participation. The primary endpoint was the magnitude of the (CP) measured by the tool grading scale of chronic pain (EGDC), while as secondary were considered the cardiovascular risk factors, catastrophism, kinesiofobia, disabled by back pain, quality of life, anxiety and depression and the (FA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain more than 3 months
* Age over 18 years old
* Low or Medium Cardiovascular Risk

Exclusion Criteria:

* Cardiovascular Risk Factors ≥ 5
* Quirurgic procedures at spine last 10 years
* Past of Cancer, or Fibromialgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Severity of Chronic Pain | 1 month
  Graded Chronic Pain Scale

SECONDARY OUTCOMES:
Amount of Physical Activity | 1 month
  International Physical Activity Questionnaire
Kinesiophibia | 1 month
  Tampa Scale of Kinesiophobia
Catastrophism | 1 month
  Pain Catastrophicing Scale
Cardiovascular Risk Factors | 1 month
  American College of Sports Medicine description of 8 Cardiovascular Risk Factors
Anxiety and Depression | 1 month
  Hospital Anxiety and Depression Scale
Low Back Pain Percieved Disability | 1 month
  Roland Morris Disability Questionnaire
Quality of Life | 1 month
  EuroQoL 5D- 5L

CONTACTS AND LOCATIONS:
Locations (1):
- CS Entrevías, Madrid, Madrid, Spain

REFERENCES:
- [Background] Phillips K, Clauw DJ. Central pain mechanisms in the rheumatic diseases: future directions. Arthritis Rheum. 2013 Feb;65(2):291-302. doi: 10.1002/art.37739. No abstract available. PMID 23045168
- [Background] O'Sullivan P. Diagnosis and classification of chronic low back pain disorders: maladaptive movement and motor control impairments as underlying mechanism. Man Ther. 2005 Nov;10(4):242-55. doi: 10.1016/j.math.2005.07.001. Epub 2005 Sep 9. PMID 16154380
- [Background] Gore M, Sadosky A, Stacey BR, Tai KS, Leslie D. The burden of chronic low back pain: clinical comorbidities, treatment patterns, and health care costs in usual care settings. Spine (Phila Pa 1976). 2012 May 15;37(11):E668-77. doi: 10.1097/BRS.0b013e318241e5de. PMID 22146287
- [Background] Philips HC. Avoidance behaviour and its role in sustaining chronic pain. Behav Res Ther. 1987;25(4):273-9. doi: 10.1016/0005-7967(87)90005-2. No abstract available. PMID 3662989
- [Background] Lethem J, Slade PD, Troup JD, Bentley G. Outline of a Fear-Avoidance Model of exaggerated pain perception--I. Behav Res Ther. 1983;21(4):401-8. doi: 10.1016/0005-7967(83)90009-8. No abstract available. PMID 6626110
- [Background] Ryan CG, Grant PM, Dall PM, Gray H, Newton M, Granat MH. Individuals with chronic low back pain have a lower level, and an altered pattern, of physical activity compared with matched controls: an observational study. Aust J Physiother. 2009;55(1):53-8. doi: 10.1016/s0004-9514(09)70061-3. PMID 19226242